CLINICAL TRIAL: NCT06922006
Title: Is Radiation Free Percutaneous Nephrolithotomy (PCNL) Feasible: A Prospective Trial
Brief Title: Feasibility of Radiation-Free Percutaneus Nephrolithotomy for Kidney Stones
Acronym: PCNL
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Roger L Sur, M.D., Professor of Urology, University of California, San Diego
Other Study IDs: IRB#180946
Record Dates: First submitted 2025-03-27; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Kidney Stones
Keywords: PCNL
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Radiation-free PCNL: Cases that were done using ultrasound as the only imaging modality during the entire procedure.
  Interventions: Procedure: Percutaneus nephrolithotomy (PCNL)
- Fluoroscopy-guided PCNL: Traditional PCNL's that were planned and performed with fluoroscopy.
  Interventions: Procedure: Percutaneus nephrolithotomy (PCNL)
- Converted from radiation-free to fluoroscopy-guided PCNL: Cases that were planned to be done with ultrasound but that ended up having to use fluoroscopy.
  Interventions: Procedure: Percutaneus nephrolithotomy (PCNL)

INTERVENTIONS:
Procedure: Percutaneus nephrolithotomy (PCNL) — Percutaneus nephrolithotomy (PCNL) for removal of large kidney stones

SUMMARY:
The goal of this observational study is to investigate the feasibility of ultrasound-guided percutaneus nephrolithotomy in patients with kidney stones. The main question's it aims to answer are:

Does the use of ultrasound in percutaneus nephrolithotomy affect stone free rates, defined by no stone or stone <2mm, on follow up visit?

Does the use of ultrasound in percutaneus nephrolithotomy affect complication rates, categorized by Clavien system?

Researchers will compare ultrasound-guided percutaneus nephrolithotomy to traditional nephrolithotomy using fluoroscopy to see if outcomes differ.

Participants will be chosen for any of the above interventions at surgeon's discretion.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is a minimally invasive procedure for removal of kidney stones that has traditionally been done using fluoroscopy for guidance. This study aims to explore if PCNL can be done safely using ultrasound as a replacement for fluoroscopy to decrease radiation exposure.

This study is a prospective cohort comparing subjects that undergoes radiation free and non-radiation free PCNLs performed by a single surgeon at UCSD Health. All cases are evaluated for ultrasound feasibility, and some have to be converted to fluoroscopy at surgeon's discretion. Information about the risks of the procedure including bleeding, infection, incomplete stone removal and injury to the kidney is given to each participant. All surgeries are performed by an experienced urologist with a history of successful ultrasonography interpretation and fluoroscopy is always accessible in the OR in case ultrasonography would not offer good enough imaging quality for the procedure to be completed in a safe and successful manner. The study does not affect the choice of imaging modality used for individual procedures but only looks at characteristics and outcomes of already performed surgeries.

Subjects are selected from the schedule in Epic and divided into three groups, radiation free PCNLs, converted cases and planned PCNLs with fluoroscopy based on information provided in the operative note from each procedure. All subjects that appear on the schedule are included in this study. Data is collected from a US electronic medical record system (Epic), using an online database tool, RedCap. The data consists of 15 cases that have undergone radiation free PCNL, 15 cases that were converted to fluoroscopy, 32 cases that were planned and performed with fluoroscopy. 5 operations had to be aborted. Data is divided into patient demographics (age, gender, ethnicity, BMI, past medical history, anticoagulants), pre-operative data (ASA class, pre-op tubes, laterality, total stone burden, number of stones, stone location, pre-op urine culture, reason for radiation or radiation-free procedure), operative data (imaging modality, access location, number of access attempts, tract dilation size, end of tube case, estimated blood loss, end of case residual stones, total time in operating room (OR), total time under fluoroscopy) and postoperative data (admissions, hospital length of stay, inpatient course, discharge antibiotics, 30 day complications, post-op imaging, post-op stone size, need for additional procedure, post-op creatinine levels and GFR).

ELIGIBILITY:
Inclusion Criteria:

Scheduled percutaneus nephrolithotomy by Dr. Roger Sur between 2022 and 2025 at UCSD Hillcrest.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General population with kidney stones larger than 20mm.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Stone free rates | 4-6 weeks after surgery.
  The rate of patients with no stone, or <2mm stone on follow up visit.

SECONDARY OUTCOMES:
Complication rates | From date of surgery to 30 days post surgery.
  Rate of complications defined by Clavien stage 1-5.
ED visits | From surgery to 30 days after surgery.
  Rate of patients that had to visit the emergency departent after the surgery.
Re-admission rates | From surgery to 30 days after surgery.
  Rate of patients that had to be re-admitted after the surgery.
Required additional procedure after PCNL. | From surgery to 30 days after surgery.
  Rate of patients that had to be planned for additional procedure after the surgery.
End of case residual stone prescense. | At the end of surgery (In the operating room).
  Rate of patients that had a residual stone visible after the procedure.
Post-operative stone size | 4-6 weeks after surgery.
  Size of kidney stone on follow up visit after the surgery.
Hospital length of stay. | From surgery to 4-6 weeks after surgey.
  Amount of days spent in hospital post-operatively.
Post-operative outpatient creatinine levels | From 30 days after surgery to next available creatinine level available in medical records.
  Creatinine levels.
Post-operative glomerulal filtration rate (GFR) | From 30 days after surgery to next available creatinine level available in medical records.
  Glomerulal filtration rate (GFR) as an indicator of kidney function post-operatively.
Estimated blood loss | From the time of incision to the time of closure.
  Amount of blood loss the patient had during the surgery.
Total OR time | From when the patient enters the operating room until the patient leaves the operating room.
  Time spent in the operating room
Incision to close time | From the first incision until closure of the last incision.
  Time spent operating.

CONTACTS AND LOCATIONS:
Overall Officials: Roger L Sur, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, Hillcrest, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided